CLINICAL TRIAL: NCT03036449
Title: Efficacy of Tools Associated With a Multifaceted Education Intervention Directed to Health Professionals to Reduce Medication Preparation and Administration Error Rates in Neonatal Intensive Care Units
Brief Title: Efficacy of a Multifaceted Intervention to Reduce Medication Administration Errors in Neonatal Intensive Care Units
Acronym: OREANE
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2014/38
Record Dates: First submitted 2016-12-23; First posted 2017-01-30 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Neonatal Intensive Care
Keywords: Medication errors; Patient safety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- A: Group A: Phase 1: Observations (Baseline rate of errors); Phase 2: Main Educational program; Phase 3: Observations; Phase 4: Maintenance Educational program; Phase 5: Observations; Phase 6: Maintenance Educational program; Phase 7: Observations; Phase 8: Maintenance Educational program; Phase 9: Observations.
  Interventions: Behavioral: Education program for NICU caregivers.
- B: Group B: Phase 1: Observations (Baseline rate of errors); Phase 2: No intervention; Phase 3: Observations (Baseline rate of errors); Phase 4: Main Educational program; Phase 5: Observations; Phase 6: Maintenance Educational program; Phase 7: Observations; Phase 8: Maintenance Educational program; Phase 9: Observations.
  Interventions: Behavioral: Education program for NICU caregivers.
- C: Group C: Phase 1: Observations (Baseline rate of errors); Phase 2: No intervention; Phase 3: Observations (Baseline rate of errors); Phase 4: No intervention; Phase 5: Observations (Baseline rate of errors); Phase 6: Main educational program; Phase 7: Observations; Phase 8: Maintenance educational program; Phase 9: Observations.
  Interventions: Behavioral: Education program for NICU caregivers.

INTERVENTIONS:
Behavioral: Education program for NICU caregivers. — Intervention includes a main initial educational program, maintenance education programs and tools supply
  - Main educational program will include 9 hours of courses into NICU (1 hour each week) and @ learning modules validation.
  Topics: Main causes of medication errors, How to analyse retrospectively medication errors, Strategies to reduce medication errors, How to improve communication between health professional; Task interruption; Standardisation of preparation…..
  * Maintenance education program will return on specific topics of main program and will be fitted to each NICU needs.
  * Examples of Tools: check lists, medication neonatal formulary, "Sound alike" and "Look alike" drug lists…

SUMMARY:
The purpose of this study is to determine whether an educational program for caregivers associated with convenient tools is effective to reduce medication preparation and administration errors in the Neonatal Intensive Care Units (NICU).

DETAILED DESCRIPTION:
Medication errors are frequent in neonatal intensive care units and consequences are more severe than in adults. Although errors happen in each step of medication management process, a large proportion of errors occur during medication preparation and administration.

This study will test the hypothesis that rates of medication errors during preparation and administration will be reduced by implementing an education program for NICU caregivers (Nurses) and providing convenient tools.

The trial has a stepped wedge design, in which the NICU's from three hospitals in France will be randomized (Group A, B and C) to the timing of implementation of the educational intervention.

According to the allocation (Group A, B or C), the education intervention will include a complete main program of nine weeks and one to three maintenance educational periods.

Medication administration errors rates will be measured before (baseline measurements) and after each educational interventions (main or maintenance interventions).

Errors will be identified by direct observations of nurse's acts by external observers.

ELIGIBILITY:
Inclusion Criteria:

* All nurses working in the intensive care units in the day time.

Exclusion Criteria:

* Nurses working as a float or pool nurses.
* Nurses working at night.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients less than 2 years old, hospitalized in the intensive care during the observation periods and receiving drugs.
Sampling Method: Non-Probability Sample
Enrollment: 5143 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2019-03-17 (Actual); Study Completion 2019-03-17 (Actual)

PRIMARY OUTCOMES:
Medication administration error rates in the patients | Baseline and up to 49 weeks
  Assessment of the efficacy of the intervention on reducing the rates of medication administration errors.
  Error rate: Number of identified errors/Number of observed acts of administration*100, measured by direct observation of nurse's acts by specifically trained external observers.

SECONDARY OUTCOMES:
Levels of safety culture among the caregivers (Nurses) | Baseline and up to 49 weeks
  Assessment of the effectiveness of the educational intervention on increasing safety culture measured using Hospital Survey on patient safety.
Levels of medication errors reported by caregivers. | Baseline and up to 49 weeks
  Assessment of the efficacy of the educational intervention to increase voluntary reporting of medication errors by caregivers.
Acceptance of the educational program | Baseline and up to 49 weeks
  Assessment of acceptance by satisfaction questionnaire

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Service de pédiatrie - Hôpital Pellegrin, Bordeaux
  - CHU Côte de Nacre, Caen
  - CHU de Rouen, Rouen